CLINICAL TRIAL: NCT00100724
Title: A Phase 2 Multi-Center, Randomized Dose-Finding Trial of rPA-102 Vaccine in Healthy Adult Volunteers
Brief Title: Trial of rPA-102 Vaccine in Healthy Adult Volunteers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: VaxGen (Industry)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH); Centers for Disease Control and Prevention (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VAX006
Record Dates: First submitted 2005-01-05; First posted 2005-01-06 (Estimated); Last update posted 2006-01-12 (Estimated); Status verified 2006-01

CONDITIONS: Anthrax
Keywords: Anthrax; rPA102; vaccine
MeSH Terms: conditions — Anthrax

INTERVENTIONS:
Biological: rPA102

SUMMARY:
The purpose of this study is to assess the safety and immunogenicity of rPA102 vaccine given intramuscularly at 0 and 4 weeks over 2 dose ranges and 4 adjuvant levels.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the study and give written informed consent. A signed informed consent must be in place before the initiation of any study interventions.
* Healthy male or female aged 18-55 years old (inclusive) without significant physical or clinical laboratory abnormalities.
* Two intact upper arms with sufficient intramuscular (IM) tissue in the deltoid region for vaccine administration.
* For females, negative serum pregnancy test at screening and agreement to use adequate birth control during the first 2 months of the study.
* Willingness and ability to return for all follow-up visits and blood draws for the duration of the study.
* Willingness to complete the Volunteer Diary and to report concomitant medications and adverse events (AEs) to the study site monitors during the study period.

Exclusion Criteria:

* Prior history of, or known exposure to any form of B. anthracis or any anthrax immunization.
* Member of the Armed Services (Active Duty or Reserve) since 1990, with history of previous anthrax vaccination.
* Employment in an industry involved in contact with ruminant animals, veterinary sciences, or other exposure to B. anthracis, or emergency first responders.
* Expected to be noncompliant with study visits or planning to move within 12 months.
* Body mass index of >35 or <19.
* Known allergy to aluminum hydroxide, kanamycin, or any other aminoglycoside antibiotics (such as gentamicin).
* Pregnancy (positive urine pregnancy test within 24 hours prior to vaccination), or lactation.
* HIV positive (by history or screening ELISA).
* Hepatitis B or C positive (by history or screening HBsAg/anti-HCV ELISA).
* Active or past internal organ, hematologic malignancy, or metastatic cutaneous malignancy.
* History of, or current autoimmune disease, including but not limited to systemic lupus erythematosus, scleroderma, and polyarteritis.
* Immunodeficiency or unstable medical condition as determined by baseline medical history, physical exam, and laboratory assessment.
* Received or plans to receive licensed live vaccines within 30 days of study vaccination.
* Received or plans to receive licensed killed vaccines within 14 days of study vaccination.
* Received or plans to receive immunoglobulin or other blood products within 60 days of study vaccination.
* Received or plans to receive experimental drugs/vaccines within 30 days prior to, and for the duration of the study.
* Received or plans to receive systemic immunosuppressive therapy, radiation therapy, or high-dose inhaled steroids within 30 days of study vaccination.
* Use of systemic chemotheraphy within 5 years prior to study.
* History of Guillain-Barre Syndrome.

In addition to the conditions listed above, the following may qualify as a reason to exclude a volunteer from the study: fever along with moderate or serious illness within 3 days of vaccination or any condition that, in the opinion of the investigator, would render vaccination unsafe or would interfere with the study evaluations. Pending resolution of these symptoms, a volunteer may be reconsidered for vaccination.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 480
Dates: Start 2004-04; Study Completion 2005-07

PRIMARY OUTCOMES:
Safety and immune response to vaccine.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - UCLA Ctr for Vaccine Research, LA Biomedical Research Institute, Torrance, California
  - Emory Children's Clinic, Pediatric Infectious Disease, Atlanta, Georgia
  - University of Kentucky, Markey Cancer Center, Lexington, Kentucky
  - Johns Hopkins University, Bloomberg School of Public Health, Baltimore, Maryland
  - Mayo Clinic College of Medicine, Rochester, Minnesota
  - St. Louis University, SoLUtions, St Louis, Missouri
  - Infectious Disease Unit, University of Rochester Medical Center, Rochester, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Pediatric Clinical Trials Int'l, Inc. (PCTI), Columbus, Ohio
  - Primary Physicians Research, Inc., Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - University of Vermont College of Medicine, Vermont Vaccine Evaluation Center, Burlington, Vermont